CLINICAL TRIAL: NCT05989789
Title: Radioactive Seed-guided Resection of Cholangiocellular Carcinoma in Cirrhotic Patients - Report of Two Cases
Brief Title: Radioactive Seed-guided Resection of Cholangiocellular Carcinoma in Cirrhotic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clarunis - Universitäres Bauchzentrum Basel (Other)
Responsible Party: Principal Investigator, Savas Soysal, Principal Investigator, Clarunis - Universitäres Bauchzentrum Basel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019_02118
Record Dates: First submitted 2023-06-26; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Liver Cancer; Liver Cirrhosis
MeSH Terms: conditions — Liver Neoplasms; Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radioactive seed-guided resection of cholangiocellular carcinoma in cirrhotic patients (Other): Detection of cholangiocellular and hepatocellular carcinomas can be challenging in both radiologic imaging and during surgical resection. Therefore, radioactive seed-guided resection of these tumors, analogously to breast cancer, could be an interesting approach.
  This report emphasizes the difficulties, which surgeons and radiologists may face in tumor entities that are difficult to identify both macroscopically, by palpation and intraoperative imaging techniques. It also highlights the successful adaption of a procedure commonly used for breast cancer surgery for liver surgery
  Interventions: Device: Radioactive Seed Implantation

INTERVENTIONS:
Device: Radioactive Seed Implantation — In patients where initially the tumour lesion could not be identified, a radioactive seed was implanted and intraoperatively detected with a geiger counter sonde.

SUMMARY:
Detection of cholangiocellular and hepatocellular carcinomas can be challenging in both radiologic imaging and during surgical resection. Therefore, radioactive seed-guided resection of these tumors, analogously to breast cancer, could be an interesting approach. The investigators present two cases of cirrhotic patients where this method of tumor labelling was used.

DETAILED DESCRIPTION:
The investigators selected two cases of patients with liver cirrhosis where seed-guided liver resection was used. Seed-guided resection is procedure that is usually commonly used in breast cancer surgery but so far not in liver surgery.

This report emphasizes the difficulties, which surgeons and radiologists may face in tumor entities that are difficult to identify both macroscopically, by palpation and intraoperative imaging techniques.

The first case was a patient suffering from suspected hepatocellular carcinoma with the background of alcoholic liver cirrhosis. This patient already underwent liver surgery to remove the suspected tumour but the lesion could not be removed correctly as identification was not possible neither with palpation nor with the help of intraoperative ultrasound. For this reason, the patient was selected for seed-guided resection.

The second patient, who presented nine months after the first one, presented with the suspicion of cirrhosis, two lesion small in size and in a surgically difficult localization. Therefore, the patient was selected for seed-guided resection.

ELIGIBILITY:
Inclusion Criteria:

* suspect cancerous liver lesion
* fit for surgery

Exclusion Criteria:

* emergency surgery
* age under 18

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-03-27 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
R0-Resection according to the tumour classification system | 1 week after operation
  Removal of the tumour in healthy tissue, which means that microscopically no tumour tissue is detectable in the resection margin of the removed tissue.
  This is always examined by a trained pathologist.
Procedure-Safety (No residual source of radiation) | 1 Day
  Complete seed extraction was confirmed intraoperatively by specimen radiography immediately after tissue removal and by ensuring that no residual source of radiation is traceable in the patient with the gamma probe system.

SECONDARY OUTCOMES:
Number of patients without side effects | 6 months
  Clinical follow up of the patients to ensure that there are no side effects from implanting the Seed in the liver

CONTACTS AND LOCATIONS:
Overall Officials: Savas D Soysal, Professor, Principal Investigator — Clarunis Basel
Locations (1):
- University hospital, Basel, Switzerland